CLINICAL TRIAL: NCT04404556
Title: Diabetes Journey: An Intervention to Improve Adherence Barriers for Adolescents With Type 1 Diabetes
Brief Title: Diabetes Journey: An Adolescent Adherence Barriers Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: University of Florida (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-0162; R01DK121295 (NIH)
Record Dates: First submitted 2020-05-19; First posted 2020-05-27 (Actual); Results first posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-06

CONDITIONS: Type 1 Diabetes; Adherence, Patient
Keywords: Adolescent; mHealth; executive functioning skills; adherence barriers
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Patient Compliance

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of two conditions: 1) Diabetes Journey or 2) Enhanced Standard of Care.
Who Masked: Care Provider
Masking Description: Outcome measures are patient-reported and thus masking will not occur at the level of participant, investigator or outcomes assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetes Journey (Experimental): Diabetes Journey is a web-based intervention to address key adherence barriers. Participants randomized to this arm will first receive the mandatory Introduction and Problem-Solving Module. Based on their elevations on the Barriers to Diabetes Adherence measure, participants will receive up to 7 modules in total. Participants will navigate through the web-based theme park map and complete modules independently and then will have accompanying Zoom telehealth sessions with a therapist.
  Interventions: Behavioral: Diabetes Journey
- Enhanced Standard of Care (Active Comparator): Participants randomized to Enhanced Standard of Care will receive general education via the T1DToolkit website, as well as 4 phone calls with certified diabetes educators (CDEs) from each site across 12-weeks. Content to address adherence barriers were modified and or newly developed for the Enhanced Standard of Care group via the T1DToolkit website.
  Interventions: Behavioral: Enhanced Standard of Care

INTERVENTIONS:
Behavioral: Diabetes Journey — Web-based telehealth intervention focused on adherence barriers and problem-solving
  Other Names: mHealth problem-solving adherence barriers intervention
  Arms: Diabetes Journey
Behavioral: Enhanced Standard of Care — General education via the T1DToolkit website, as well as 4 phone calls with certified diabetes educators (CDEs) will be provided.
  Other Names: t1dtoolkit
  Arms: Enhanced Standard of Care

SUMMARY:
The purpose of this study is to examine the feasibility, acceptability, and preliminary efficacy of a web-based intervention addressing adherence barriers in adolescents with T1D.

DETAILED DESCRIPTION:
Type 1 diabetes (T1D) treatment adherence is complex and involves glucose monitoring, counting carbohydrates, and intensive insulin delivery via injections or insulin pump in response to food intake, exercise, and illness to achieve near-normal blood glucose levels. Evidence demonstrates that adhering to T1D treatment is challenging, especially during adolescence. Non-adherence leads to suboptimal glycemic levels that severely compromise health and quality of life. Suboptimal adherence to T1D treatment regimen is common in >50% of adolescents and directly related to suboptimal glycemic control, increased risk of hospitalizations for diabetic ketoacidosis, and decreased health-related quality of life (HRQOL). The maximum benefits of current diabetes technology are limited by the knowledge, skills, adherence barriers, and non-adherence behaviors.10-14 Ultimately, adolescents have to overcome these barriers in order to benefit from technological advances. Thus, there is a clear need for behaviorally focused interventions to identify and reduce adherence barriers. The overall objective of this study is to identify adolescents with elevated adherence barriers and provide novel tailored mHealth intervention (Diabetes Journey) targeting these barriers. This study is two phases and includes a small pilot of up to 12 adolescents with type 1 diabetes (Phase 1) and a randomized controlled clinical trial (Phase 2). The randomized controlled clinical trial will examine feasibility, acceptability and preliminary efficacy of Diabetes Journey versus enhanced standard of care (control group) in approximately 256 adolescents with type 1 diabetes. Primary and secondary outcomes include adherence barriers, adherence, health-related quality of life and A1C. Satisfaction and acceptability will also be examined. Mediators and moderators will include executive functioning, diabetes distress, family conflict, depressive symptoms, fear of hypoglycemia and sleep.

ELIGIBILITY:
Inclusion Criteria

* T1D diagnosis >1 year
* Adolescents with T1D ages 13-17
* Elevations on the Barriers to Diabetes Adherence questionnaire (scores of ≥3 of 53 for the Stress/Burnout and/or Time Pressure/Planning subscales) based on their previous clinic visit scores
* Ability to read/speak English (all measures are in English)

Exclusion Criteria

* Diagnosis of significant developmental disorders (e.g., autism spectrum disorder, moderate/severe developmental or intellectual disability)
* Comorbid medical diagnoses (e.g., cystic fibrosis, asthma) with the exception of endocrine disorders (e.g., Celiac disease, thyroid)
* No use of/plans to use non-insulin medication for blood glucose control

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 195 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Florida, Gainesville, Florida
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: Yes
The NIDDK Data Repository will serve as the primary data repository for the current proposal.
Time Frame: The NIDDK Data Repository will serve as the primary data repository for the current proposal. In addition, data sets may also be distributed via clinicaltrials.gov. Should individuals or organizations request the dataset directly from the principal investigators, those requests will be directed to the NIDDK Data repository to retrieve the data.
  Per NIDDK guidelines on resource sharing for intervention studies, baseline data will be shared within 2 years after study recruitment is complete or within six months of the publication date of the baseline data, whichever comes first. An analytic dataset for the baseline publication will be provided within 6 months of the publication date (when the publication appears online).
Access Criteria: The investigators agree that they will identify where the data will be available and how to access the data in any publications and presentations that the investigators author or co-author about these data, as well as acknowledge the repository and funding source in any publications and presentations. Since the investigators will be using the NIDDK Data Repository, this repository has policies and procedures in place that will provide data access to qualified researchers, fully consistent with NIH data sharing policies and applicable laws and regulations.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After participants were consented, there was a screening process. If participants were elevated on the BDA, they were eligible to be randomized. If they were not elevated, they screen failed. Of the 195 participants who were consented, n=13 screen failed and additional n=20 withdrew prior to randomization. Thus, only n=162 were randomized.
Period: Intervention
Arm/Group | Diabetes Journey | Enhanced Standard of Care
Started | 97 | 65
Completed | 80 | 61
Not Completed | 17 | 4
Not completed — Withdrawal by Subject | 15 | 3
Not completed — Did not complete all intervention sessions | 2 | 1
Period: Post-Intervention
Arm/Group | Diabetes Journey | Enhanced Standard of Care
Started | 82 | 62
Completed | 81 | 60
Not Completed | 1 | 2
Not completed — Missing Data | 1 | 2
Period: Follow-up 1
Arm/Group | Diabetes Journey | Enhanced Standard of Care
Started | 81 | 62
Completed | 72 | 54
Not Completed | 9 | 8
Not completed — Withdrawal by Subject | 5 | 1
Not completed — Missing Data | 4 | 7
Period: Follow-up 2
Arm/Group | Diabetes Journey | Enhanced Standard of Care
Started | 63 | 50
Completed | 56 | 44
Not Completed | 7 | 6
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Missing Data | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diabetes Journey | Enhanced Standard of Care | Total
Number analyzed (Participants) | 97 | 65 | 162
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.82 (1.49) | 14.74 (1.72) | 14.79 (1.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 37 | 93
  Male | 41 | 28 | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 8 | 14
  Not Hispanic or Latino | 91 | 57 | 148
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 3 | 8
  White | 86 | 56 | 142
  More than one race | 5 | 5 | 10
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Barriers to Diabetes Adherence Questionnaire-Youth Report Stress/Burnout Subscale
Description: Stress and Burnout Scale - assesses frustration and feeling burned out by diabetes and its management. Score range from 1-5, with higher scores representing greater barriers.
Time Frame: 6-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Diabetes Journey | Enhanced Standard of Care
Number analyzed (Participants) | 72 | 54
score on a scale | 2.36 (0.90) | 2.31 (1.05)

2. Primary Outcome: Barriers to Diabetes Adherence Questionnaire - Youth Report Time Pressure/Planning Subscale
Description: Time Pressure and Planning Subscale - assesses the time and energy it takes to plan for diabetes self-management, including carrying supplies and making management decisions. Score range from 1-5, with higher scores representing greater barriers.
Time Frame: 6-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Diabetes Journey | Enhanced Standard of Care
Number analyzed (Participants) | 72 | 54
score on a scale | 1.92 (0.58) | 2.03 (0.89)

3. Secondary Outcome: Hemoglobin A1C
Description: A blood test that measures the average blood sugar levels over the past two to three months.
Time Frame: 6-month follow-up
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Diabetes Journey | Enhanced Standard of Care
Number analyzed (Participants) | 63 | 49
percentage of glycosylated hemoglobin | 8.06 (1.72) | 7.98 (1.67)

4. Secondary Outcome: Type 1 Diabetes and Life -Youth Report
Description: Total Quality of Life Scores range from 0-100, with higher scores indicating better quality of life
Time Frame: 6-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Diabetes Journey | Enhanced Standard of Care
Number analyzed (Participants) | 65 | 50
score on a scale | 65.84 (14.71) | 65.82 (18.32)

5. Secondary Outcome: Adherence for Continuous Glucose Monitors
Description: % Time in Range for those on continuous glucose monitors.
Time Frame: 6-month follow-up
Reporting Status: Not Posted

6. Secondary Outcome: Adherence
Description: # blood glucose checks per day
Time Frame: 6-month follow-up
Reporting Status: Not Posted

7. Secondary Outcome: Adherence for Insulin Pump Users
Description: # carbohydrate entries per day for insulin pump users
Time Frame: 6-month follow-up
Reporting Status: Not Posted

8. Secondary Outcome: Adherence to Insulin Boluses
Description: The average of the frequency of insulin boluses delivered per day
Time Frame: 6-month follow-up
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: ~9 months
Arm/Group | Diabetes Journey | Enhanced Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/97 | 0/65
Serious Adverse Events (participants affected / at risk) | 0/97 | 1/65
Other Adverse Events (participants affected / at risk) | 50/97 | 39/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diabetes Journey (N=97) | Enhanced Standard of Care (N=65)
Increased suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) — Increased frequency of suicidal ideation which involved psychiatric hospitalization
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diabetes Journey (N=97) | Enhanced Standard of Care (N=65)
Psychological Complications (Psychiatric disorders) | 45 (73) | 36 (54) — Elevations on the PHQ-8, symptoms of distress, depression, anxiety, and suicidal ideation
Medical complications not related to type 1 diabetes (Injury, poisoning and procedural complications) | 15 (17) | 9 (10) — injuries, back pain, dental abcess, broken bones, viral illness, otitis externa
Medical complications related to type 1 diabetes (Endocrine disorders) | 13 (15) | 4 (5) — DKA, accidental insulin overdose, high blood glucuse, hyperglycemia, hypoglycema, ketonuria, cellulitis
Social complication (Social circumstances) | 1 (1) | 0 (0) — Medical Neglect reported to and investigated by DCFS
Regulatory Issue (Investigations) | 0 (0) | 1 (1) — PHI Breach and possible breach

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-06-08): https://cdn.clinicaltrials.gov/large-docs/56/NCT04404556/Prot_001.pdf
  • Statistical Analysis Plan (2024-11-21): https://cdn.clinicaltrials.gov/large-docs/56/NCT04404556/SAP_002.pdf
  • Informed Consent Form (2023-06-20): https://cdn.clinicaltrials.gov/large-docs/56/NCT04404556/ICF_000.pdf